CLINICAL TRIAL: NCT06695468
Title: Efficacy and Safety of Adding Dexmedetomidine to Levobupivacaine in Rectus Sheath Block Compared to Quadratus Lumborum Block in Patients Undergoing Lower Abdominal Cancer Surgery: a Randomized Clinical Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerollos Ibrahim Gayed Ibrahim, resident doctor at Anaesthesia, I.C.U and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dexmedetomidine QLB
Record Dates: First submitted 2024-11-17; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Abdominal Cancer Surgery
Keywords: Quadratus Lumborum Block; dexmedetomidine; Levobupivacaine; Rectus sheath block
MeSH Terms: interventions — Levobupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer-generated database of random numbers will be used to randomly assign patients into two groups in a 1:1 ratio. The randomization will be carried out using a numbered, opaque, and sealed envelope.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Quadratus lumborum block (QLB group) (Experimental): patients will receive bilateral QLB with a 40-ml mixture of 20 ml of 0.5% levobupivacaine diluted with 20 ml of 0.9% N.S. (20 ml to be injected on each side).
  Interventions: Drug: Levobupivacaine
- Rectus sheath block (RSB group) (Experimental): patients will receive bilateral RSB with a 60 ml mixture of 1.5 mic/kg dexmedetomidine added to 30 ml of 0.5% levobupivacaine diluted with 30 ml of 0.9% N.S. (30 ml to be administered on each side, divided into 15 ml for the upper segment and 15 ml for the lower segment).
  Interventions: Drug: Levobupivacaine + Dexmedetomidine

INTERVENTIONS:
Drug: Levobupivacaine — 40-ml mixture of 20 ml of 0.5% levobupivacaine diluted with 20 ml of 0.9% N.S. (20 ml to be injected on each side
  Arms: Quadratus lumborum block (QLB group)
Drug: Levobupivacaine + Dexmedetomidine — 60 ml mixture of 1.5 mic/kg dexmedetomidine added to 30 ml of 0.5% levobupivacaine diluted with 30 ml of 0.9% N.S. (30 ml to be administered on each side, divided into 15 ml for the upper segment and 15 ml for the lower segment).
  Arms: Rectus sheath block (RSB group)

SUMMARY:
Surgical trauma activates numerous receptors leading to severe postoperative pain. Seventy to seventy-five percent of the pain is somatic, originating from the anterior abdominal wall, and it often persists for 72 hours after open surgery. The objective of this study is to compare the efficacy and safety of adding dexmedetomidine to Levobupivacaine in rectus sheath block with quadrates lumborum block in patients undergoing lower abdominal cancer surgeries.

DETAILED DESCRIPTION:
Postoperative pain may cause tachycardia, hypertension, increased cardiac work, nausea, vomiting and ileus. Also, if it is inadequately managed it may lead to hazardous cardiovascular effects, pulmonary dysfunction, immune system, neuro-endocrine and metabolic effects, gastrointestinal- urinary- and cognitive dysfunction and also have psychological, economic and social adverse effects. Therefore, effective pain management is a priority of care and a patient's right.

The American Society of Anesthesiologists recommends use of multimodal pain regimens to minimize opioid use and improve pain control . Opioids are still the go-to medication for treating visceral pain, but they are ineffective against somatic discomfort. An effective Multimodal pain management protocol uses combinations of opioid prescriptions, nonopioid prescription, regional and local anesthesia, and nonpharmacological therapy . To mitigate the adverse consequences of opioid overconsumption, peripheral and regional anesthetic blocks were implemented. The Quadratus lumborum block is one of the perioperative pain management procedures that is administered to patients of all ages who are undergoing abdominal surgery . Nevertheless, there is persistent disagreement regarding the optimal method of administering the block due to the ambiguous mechanisms that are responsible for its effects.

We sought an alternative, such as the Rectus sheath block, to prevent postoperative somatic pain, due to the potential complications of the QLB technique, including retroperitoneal hemorrhage, abscess, and pleural injury . The block was not frequently applied, or insufficient blocks could not be achieved primarily with a single injection method prior to taking advantage of ultrasonography. This was due to the proximity of medicated zones and vital organs, as well as the coherent and thin muscle layers. Currently, this approach is being implemented with catheter placement in the rectus sheath, ultrasonography guidance, and a single injection .

At present, several adjuvants have been added to local anesthetics used in peripheral and regional blocks to decrease the dosage of local anesthetic and enhance its effectiveness . Dexmedetomidine is an adjuvant that acts as a selective alpha two adrenoreceptor stimulating agent. This medication induces drowsiness, analgesia, sympatholysis, and anxiolysis in a dose-dependent manner, without causing significant respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients subjected to major lower abdominal cancer surgeries.
2. The enrolled age will be from 18 years to 70 years
3. ASA I-III and NYHA I-III.

Exclusion Criteria:

1. ASA physical status >III and NYHA>III
2. Patient refusal
3. Body mass index >40 kg/m2
4. Preoperative opioid consumption
5. Infection at the incision site
6. A history of hematological disorders or coagulation abnormality
7. Previous abdominal surgeries, severe hepatic or renal impairment
8. Pregnant women

10- Hypersensitivity to any of used drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 24 hours
  measured by VAS immediately postoperatively, then at 2-, 4-, 6-, 8-, 12-, 18-, 24-hours after surgery.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zheng Y, Cui S, Liu Y, Zhang J, Zhang W, Zhang J, Gu X, Ma Z. Dexmedetomidine prevents remifentanil-induced postoperative hyperalgesia and decreases spinal tyrosine phosphorylation of N-methyl-d-aspartate receptor 2B subunit. Brain Res Bull. 2012 Mar 10;87(4-5):427-31. doi: 10.1016/j.brainresbull.2012.01.009. Epub 2012 Jan 25. PMID 22301064
- [Background] Moen V, Dahlgren N, Irestedt L. Severe neurological complications after central neuraxial blockades in Sweden 1990-1999. Anesthesiology. 2004 Oct;101(4):950-9. doi: 10.1097/00000542-200410000-00021. PMID 15448529
- [Background] Okmen K, Metin Okmen B, Topal S. Ultrasound-guided posterior quadratus lumborum block for postoperative pain after laparoscopic cholecystectomy: A randomized controlled double blind study. J Clin Anesth. 2018 Sep;49:112-117. doi: 10.1016/j.jclinane.2018.06.027. Epub 2018 Jun 18. PMID 29929169